CLINICAL TRIAL: NCT00765960
Title: Evaluation of Outcomes Using the Amo Advanced CustomVue Ilasik Procedure
Acronym: iLASIK
Status: Withdrawn | Type: Observational
Why Stopped: Prinicipal Investigator separating employment from University.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kerry D. Solomon, Magill Research Center
Other Study IDs: MRC 08-002; 18294 (Other: Medical University of SC)
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2010-10

CONDITIONS: Myopia; Hyperopia
Keywords: Vision
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the efficacy, predictability and safety of the Advanced CustomVue™ iLASIK procedure (WaveScan WaveFront® System, STAR S4 IR™ Excimer Laser System and IntraLase™ FS System).

DETAILED DESCRIPTION:
Laser in situ keratomileusis (LASIK) surgery has been performed worldwide since 1990. More recently, customized corneal ablation utilizing wavefront-sensing technology to determine the optical aberration of a patient's cornea has optimized LASIK surgery results. Prior to the introduction of wavefront-guided laser vision correction, the variables used for correcting refractive errors were limited to sphere and cylinder. With the introduction of wavefront laser vision correction surgeons are now able to provide individualized laser-induced corneal tissue resection based not only on sphere and cylinder measurements, but also on an attempt to treat 3rd through 6th higher-order aberrations (HOAs) utilizing Zernike polynomial wavefront reconstructions and Fourier transformation.

Advanced Medical Optics, Inc. (AMO) has recently introduced the Advanced CustomVue™ iLASIK procedure which utilizes the WaveScan WaveFront® System, a STAR S4 IR™ Excimer Laser System and IntraLase™ FS System technology to provide the broadest range of wavefront-guided FDA approved usages and an unprecedented level of precision and accuracy for patients undergoing LASIK surgery. The procedure leverages Iris Registration, Fourier algorithms, VSS™ and VRR™ technologies and 3D ActiveTrak™ to ensure precise corneal ablation.1, 2

ELIGIBILITY:
Inclusion Criteria:Subjects MUST fulfill the following conditions to qualify for enrollment into the trial Both eyes must have a manifest refractive error from -0.50 D to -6.00 D, a cylinder component up to -3.00 D, and a maximum manifest spherical equivalent of -6.00 D.

21 years of age or older at the time of the pre-operative examination. Both eyes must have a BSCVA of 20/20 or better; Both eyes must have a minimum pupil size of at least 6.0mm in dim illumination on wavescan.

Both eyes must demonstrate refractive stability confirmed by clinical records or previous glasses. Refractive stability shall be documented by a change of less than or equal to 0.50 diopter (sphere and cylinder) at an exam at least 12 months prior to the baseline examination. The astigmatic axis must also be within 15 degrees for eyes with cylinder greater than 0.50 D.

Willing and able to comply with scheduled visits and other study procedures.

-

Exclusion Criteria:Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

Subjects who use concurrent topical or systemic medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment. Also, the use of topical or systemic corticosteroids, whether chronic or acute Subjects with a history of any of the following medical conditions, or any other condition that could affect wound healing: uncontrolled diabetes, collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

Subject must not have a history of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or with evidence of glaucoma or propensity for narrow angle glaucoma in either eye.

The subject must not have any evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.

Subjects with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.

Patients who do not achieve Iris registration at the time of their wavescan. Patients seeking monovision Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.

Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates the patient is unsuitable for the trial.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 20 patients (40 eyes) of both sexes and any race undergoing bilateral wavefront-guided LASIK will be included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Comparisons and statistical analysis will be done to determine if any statistical differences exist between preoperative and postoperative visits, and assess the efficacy, predictability and safety of the Advanced CustomVue™ iLASIK procedure. | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Professor of Ophthalmology
Locations (1):
- Magill Laser Center, Medical University of South Carolina, Charleston, South Carolina, United States